CLINICAL TRIAL: NCT05532436
Title: The Effect of Breath Exercise on Post-Operative Anxiety Level, Sleep and Recovery Quality in Laparoscopic Cholecystectomy Surgery:A Randomized Controlled Trial
Brief Title: The Effect of Breath Exercise on Patients' Post-Operative Anxiety Level, Sleep and Recovery Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Gamze BULUT, Principal İnvestigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GBULUT
Record Dates: First submitted 2022-09-05; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Cholecystectomy, Laparoscopic
Keywords: anxiety; breathing exercise; laparoscopic cholecystectomy; nurse; recovery quality; sleep quality
MeSH Terms: conditions — Anxiety Disorders; Sleep Initiation and Maintenance Disorders | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grup 1 (Experimental): One day before the operation, the participants in the experimental group were given breathing exercise training, and they were applied 5 times a day for 10 repetitions until the 30th day after the operation. Introductory Information Form, State-Trait Anxiety Scale, Visual Comparative Sleep Scale and Recovery Quality-40 Questionnaire were used to collect data 1 day before surgery, on the day of surgery, on the 1st day, 15th and 30th days after surgery.
  Interventions: Other: Breath Exercise
- Grup 2 (No Intervention): Each data collection tool was collected as in the experimental group patients, but without breathing exercises. Only routine nursing care was given to the patients in the control group. The patients in the control group were given a breathing exercise brochure/booklet when they came to the control after the postoperative 30th day, and they were shown how the breathing exercises would be done correctly.

INTERVENTIONS:
Other: Breath Exercise — It was provided by the researcher that the patients performed 5 repetitions of 10 breathing exercises every 3 hours a day, between 09:00am and 21:00pm, 1 day before the surgery, on the day of surgery and on the first day after surgery.
  Arms: Grup 1

SUMMARY:
This study was conducted to determine the effect of breath exercise on post-operative anxiety level, sleep and recovery quality after laparoscopic cholecystectomy surger. This was a randomized controlled experimental study. The sample comprised 115 patients who underwent laparoscopic cholecystectomy (control:57; experimental:58). One day before the operation, the participants in the experimental group were given breathing exercise training, and they were applied 5 times a day for 10 repetitions until the 30th day after the operation.

DETAILED DESCRIPTION:
Surgical interventions are one of the most important experiences in an individual's life and are used to improve the quality of life, to treat diseases and to improve health. Cholelithiasis is one of the most common surgical procedures that can be treated with laparoscopic cholecystectomy. Although laparoscopic surgery is a minimally invasive surgical procedure, it is expected that patients who will receive general anesthesia have an increased level of anxiety, feel pain and disrupt their sleep patterns.

The body's stress response is an expected process in coping with the problems that may develop in the post-operative period, adapting to the new situation and accelerating the recovery. However, when stressors and the response to these stressors are excessive and continuous, the healing process is adversely affected. It has been reported in the literature that patients with high anxiety levels before and after surgical intervention have a higher rate of medical complications and adversely affect wound healing.

Sleep-related problems are one of the specific consequences of the stress response to surgery.

In the literature, it has been stated that patients experience sleep problems after surgical intervention and their sleep quality is adversely affected. This situation may negatively affect the quality of life of patients, as well as increase the rate of morbidity and mortality. On the other hand, the good sleep quality of the patients affects the healing process positively and ensures early budding. In this context, well-planned patient education and nursing care management before surgery will be effective in increasing the sleep pattern and quality of patients.

Oxygenation of the traumatized tissues must be sufficient for wound healing in the postoperative incisional area. This oxygen requirement is met by effective ventilation. However, after surgery, patients have difficulty in breathing deeply due to reasons such as pain and limitation of movement. Studies have shown that the practice of planned breathing exercises reduces stress in patients in the pre- and post-operative period, provides calming, and has a positive effect on the level of pain and wound healing. In this respect, planned patient education and care to be given to patients before surgery is very effective in preventing complications related to surgical intervention.

One of the basic duties of surgical nurses is to teach and apply deep breathing and coughing exercises to the patient in pre-operative patient education. It is very important to explain the importance of these exercises to the patient and the effects of performing them at regular intervals on the quality of recovery. However, studies have drawn attention to the fact that the rates of teaching and applying deep breathing exercises to patients are not at the desired level.

Non-pharmacological applications have been widely used in recent years to improve the quality of recovery of patients after laparoscopic cholecystectomy. It has been stated in studies that deep breathing exercises, which is one of the non-pharmacological methods, reduce the anxiety level in different patient groups and increase the quality of sleep and recovery in the postoperative period. After laparoscopic cholecystectomy, the effects on many parameters such as pain, nausea-vomiting, anxiety, vital signs, early discharge, comfort, sleep and early mobilization were investigated by having patients undergo many non-pharmacological nursing practices such as cuppressor, massage, breathing exercise, music, gum chewing, and virtual reality. However, no research has been found that examines the effect of deep breathing exercise, which is planned after laparoscopic cholecystectomy, on the quality of recovery. In this context, this study was planned to determine the effect of deep breathing exercise applied to patients with laparoscopic cholecystectomy on the level of anxiety, sleep and recovery quality after surgery.

This study was conducted to determine the effect of breathing exercise on postoperative anxiety level, sleep and recovery quality in laparoscopic cholecystectomy surger. This was a randomized controlled experimental study. The sample comprised 188 patients who underwent laparoscopic cholecystectomy (control:57; experimental:58).

ELIGIBILITY:
Inclusion Criteria:

18 years and over, Having undergone laparoscopic cholecystectomy surgery with general anesthesia, They do not have physical/mental disabilities, limitations and diseases that would prevent them from doing breathing exercises (such as the use of drugs that affect breathing and requiring oxygen therapy, etc.) Cognitive level scales are suitable for application, Patients with video phones and no communication problems were included in the study.

Exclusion Criteria:

Postoperative hemodynamic values unstable, Developing any complications such as severe bleeding, nausea, vomiting after surgery, Leaving work voluntarily, Patients with acute or chronic lung disease were not included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
The State-Trait Anxiety Inventory (STAI) | 1 day before surgery
  It is a test developed by Spielberger et al. that measures state and trait anxiety levels. Its validity and reliability in Turkey was done by Oner and Le Compte. The scale consists of two parts, the 'state anxiety scale', which is created with the aim of determining the instantaneous feelings, and the 20-item 'trait anxiety scale', which was created to determine the feelings in general. It is a four degree scale ranging from 'Nothing' to 'All'. Scores range from 20 (low anxiety) to 80 (high anxiety).
The State Anxiety Inventory (SAI) | On the 1 day of surgery
  It is a test developed by Spielberger et al. that measures state and trait anxiety levels. Its validity and reliability in Turkey was done by Oner and Le Compte. The scale consists of two parts, the 'state anxiety scale', which is created with the aim of determining the instantaneous feelings. It is a four degree scale ranging from 'Nothing' to 'All'. Scores range from 20 (low anxiety) to 80 (high anxiety).
The State Anxiety Inventory (SAI) | 1st day after surgery
  It is a test developed by Spielberger et al. that measures state and trait anxiety levels. Its validity and reliability in Turkey was done by Oner and Le Compte. The scale consists of two parts, the 'state anxiety scale', which is created with the aim of determining the instantaneous feelings. It is a four degree scale ranging from 'Nothing' to 'All'. Scores range from 20 (low anxiety) to 80 (high anxiety).
The State Anxiety Inventory (SAI) | 15st day after surgery
  It is a test developed by Spielberger et al. that measures state and trait anxiety levels. Its validity and reliability in Turkey was done by Oner and Le Compte. The scale consists of two parts, the 'state anxiety scale', which is created with the aim of determining the instantaneous feelings. It is a four degree scale ranging from 'Nothing' to 'All'. Scores range from 20 (low anxiety) to 80 (high anxiety).
The State Anxiety Inventory (SAI) | 30st day after surgery
  It is a test developed by Spielberger et al. that measures state and trait anxiety levels. Its validity and reliability in Turkey was done by Oner and Le Compte. The scale consists of two parts, the 'state anxiety scale', which is created with the aim of determining the instantaneous feelings. It is a four degree scale ranging from 'Nothing' to 'All'. Scores range from 20 (low anxiety) to 80 (high anxiety).
Visual Analog Sleep Scale (VASS) | 1 day before surgery
  The VASS was developed by Verran and Snyder-Halpern in 1988 to evaluate the sleep quality of patients and healthy individuals. The Turkish validity reliability studywas performed by Çetinkaya and Karabulut in 2016. The Turkish form of the scale was created from 10 items without sub-dimensions and some items were removed, unlike the original. Each item in the scale is evaluated using the visual comparison technique on a chart from 0(at the left end) to 100 (at the right end). The Turkish form of thescale produces a score between 0 and 1000 under the title of sleepquality. The increase in the score obtained from the scale indicates that the quality of sleep decreases.
Visual Analog Sleep Scale (VASS) | On the 1 day of surgery
  The VASS was developed by Verran and Snyder-Halpern in 1988 to evaluate the sleep quality of patients and healthy individuals. The Turkish validity reliability studywas performed by Çetinkaya and Karabulut in 2016. The Turkish form of the scale was created from 10 items without sub-dimensions and some items were removed, unlike the original. Each item in the scale is evaluated using the visual comparison technique on a chart from 0(at the left end) to 100 (at the right end). The Turkish form of thescale produces a score between 0 and 1000 under the title of sleepquality. The increase in the score obtained from the scale indicates that the quality of sleep decreases.
Visual Analog Sleep Scale (VASS) | 1st day after surgery
  The VASS was developed by Verran and Snyder-Halpern in 1988 to evaluate the sleep quality of patients and healthy individuals. The Turkish validity reliability studywas performed by Çetinkaya and Karabulut in 2016. The Turkish form of the scale was created from 10 items without sub-dimensions and some items were removed, unlike the original. Each item in the scale is evaluated using the visual comparison technique on a chart from 0(at the left end) to 100 (at the right end). The Turkish form of thescale produces a score between 0 and 1000 under the title of sleepquality. The increase in the score obtained from the scale indicates that the quality of sleep decreases.
Visual Analog Sleep Scale (VASS) | 15st day after surgery
  The VASS was developed by Verran and Snyder-Halpern in 1988 to evaluate the sleep quality of patients and healthy individuals. The Turkish validity reliability studywas performed by Çetinkaya and Karabulut in 2016. The Turkish form of the scale was created from 10 items without sub-dimensions and some items were removed, unlike the original. Each item in the scale is evaluated using the visual comparison technique on a chart from 0(at the left end) to 100 (at the right end). The Turkish form of thescale produces a score between 0 and 1000 under the title of sleepquality. The increase in the score obtained from the scale indicates that the quality of sleep decreases.
Visual Analog Sleep Scale (VASS) | 30st day after surgery
  The VASS was developed by Verran and Snyder-Halpern in 1988 to evaluate the sleep quality of patients and healthy individuals. The Turkish validity reliability studywas performed by Çetinkaya and Karabulut in 2016. The Turkish form of the scale was created from 10 items without sub-dimensions and some items were removed, unlike the original. Each item in the scale is evaluated using the visual comparison technique on a chart from 0(at the left end) to 100 (at the right end). The Turkish form of thescale produces a score between 0 and 1000 under the title of sleepquality. The increase in the score obtained from the scale indicates that the quality of sleep decreases.
Quality of Recovery Scale (QoR-40) | 1 day before surgery
  The QoR-40 questionnaire, defined by Myles and colleagues in 2000, is a self-rating questionnaire used to evaluate patients' postoperative recovery quality and health status in the early postoperative stages. The QoR-40 consists of two parts, 40 items across five QoR dimensions: physical comfort (12 items), emotional state (9 items), physical independence (5 items), psychological support (7 items), and pain (7 items). Each item was rated on a five-point Likert scale, ranging from one (worst) to five (best), where 1 = none of the time, 2 = some of the time, 3 = usually, 4 = most of the time, and 5 = all the time. The total score ranges from 40 (worst recovery quality) to 200 (best recovery quality).
Quality of Recovery Scale (QoR-40) | 1st day after surgery
  The QoR-40 questionnaire, defined by Myles and colleagues in 2000, is a self-rating questionnaire used to evaluate patients' postoperative recovery quality and health status in the early postoperative stages. The QoR-40 consists of two parts, 40 items across five QoR dimensions: physical comfort (12 items), emotional state (9 items), physical independence (5 items), psychological support (7 items), and pain (7 items). Each item was rated on a five-point Likert scale, ranging from one (worst) to five (best), where 1 = none of the time, 2 = some of the time, 3 = usually, 4 = most of the time, and 5 = all the time. The total score ranges from 40 (worst recovery quality) to 200 (best recovery quality).
Quality of Recovery Scale (QoR-40) | 15st day after surgery
  The QoR-40 questionnaire, defined by Myles and colleagues in 2000, is a self-rating questionnaire used to evaluate patients' postoperative recovery quality and health status in the early postoperative stages. The QoR-40 consists of two parts, 40 items across five QoR dimensions: physical comfort (12 items), emotional state (9 items), physical independence (5 items), psychological support (7 items), and pain (7 items). Each item was rated on a five-point Likert scale, ranging from one (worst) to five (best), where 1 = none of the time, 2 = some of the time, 3 = usually, 4 = most of the time, and 5 = all the time. The total score ranges from 40 (worst recovery quality) to 200 (best recovery quality).
Quality of Recovery Scale (QoR-40) | 30st day after surgery
  The QoR-40 questionnaire, defined by Myles and colleagues in 2000, is a self-rating questionnaire used to evaluate patients' postoperative recovery quality and health status in the early postoperative stages. The QoR-40 consists of two parts, 40 items across five QoR dimensions: physical comfort (12 items), emotional state (9 items), physical independence (5 items), psychological support (7 items), and pain (7 items). Each item was rated on a five-point Likert scale, ranging from one (worst) to five (best), where 1 = none of the time, 2 = some of the time, 3 = usually, 4 = most of the time, and 5 = all the time. The total score ranges from 40 (worst recovery quality) to 200 (best recovery quality).

CONTACTS AND LOCATIONS:
Overall Officials: Gamze BULUT, Principal Investigator — Ataturk Unıversty
Locations (1):
- Gamze BULUT, Erzurum, Palandöken, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No